CLINICAL TRIAL: NCT06080074
Title: Multicenter Trial to Evaluate the Safety and Effectiveness of the Cardiohelp System for up to 30 Days of Support in Children With Severe Cardiac Failure
Brief Title: Multicenter Trial of ECMO in Children With Severe Cardiac Failure Using the Cardiohelp System
Acronym: TROLLEY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Boston Children's Hospital (Other); Duke University (Other); FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Almond, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72467
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Cardiogenic Shock; Congenital Heart Disease; Cardiomyopathies
Keywords: blood thinner; ECMO; heart failure; bivalirudin; heparin; FDA regulation; pediatric medical devices; 510k clearance
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic; Heart Defects, Congenital; Cardiomyopathies | interventions — Heparin; bivalirudin

STUDY DESIGN:
Intervention Model Description: Participants receiving ECMO with the Cardiohelp Device for severe heart failure will managed/treated according to a standardized treatment and monitoring protocol that includes anticoagulation strategy, circuit change criteria, weaning guidelines, and recording of adverse events using standardized SAE definitions adapted from the ECMO-CENTRAL guidelines.
  While the Cardiohelp device trial is a single-arm cohort study, the FDA allowed us to randomize patients to blood thinner (heparin and bivalirudin). Both blood thinners are in common use in the US--providing the FDA with safety and effectiveness data on each of the two anticoagulants in at least ~25 participants.
  Please note: Because the data fields for clinicaltrials.gov make it easier to report more robust details for a randomized clinical trial, we have chosen to report the details of the RCT in this section, understanding that the FDA clearance study is running in the background as a single arm observational study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cardiohelp device managed according to a standardized guideline using heparin anticoagulation (Experimental): Participants receiving the Cardiohelp device for severe heart failure will be managed according to a standardized treatment guideline (equipment, monitoring, etc.) where heparin is the primary blood thinner to estimate the safety and effectiveness of the device and blood thinner strategy for up to 30 days of support.
  Interventions: Device: Cardiohelp device (VA-ECMO); Drug: Heparin
- Cardiohelp device managed according to a standardized guideline using bivalirudin anticoagulation (Experimental): Participants receiving the Cardiohelp device for severe heart failure will be managed according to a standardized treatment guideline (equipment, monitoring, etc.) where bivalirudin is the primary blood thinner to estimate the safety and effectiveness of the device and blood thinner strategy for up to 30 days of support.
  Interventions: Device: Cardiohelp device (VA-ECMO); Drug: Bivalirudin

INTERVENTIONS:
Device: Cardiohelp device (VA-ECMO) — The Cardiohelp system is a compact cardiopulmonary support system used off-label for ECMO for patients with cardiac and/or respiratory failure. It is currently FDA-cleared for <6 hours of support for cardiopulmonary bypass.
Drug: Heparin — Blood thinner that works by inactivating factor Xa that is administered as a continuous intravenous infusion.
  Arms: Cardiohelp device managed according to a standardized guideline using heparin anticoagulation
Drug: Bivalirudin — Blood thinner that works by inhibiting thrombin directly that is administered as a continuous intravenous infusion.
  Arms: Cardiohelp device managed according to a standardized guideline using bivalirudin anticoagulation

SUMMARY:
There are two primary goals of this multicenter clinical trial that combines an FDA device trial and a phase II drug trial in the same study cohort. These two goals are to:

1. To evaluate the safety and effectiveness of the Cardiohelp Device for VA-ECMO (heart-lung support) for up to 30 days of support in children with severe heart failure with the goal to support its FDA clearance in children.
2. To evaluate heparin versus bivalirudin as the primary blood thinner (anticoagulant) in a randomized trial of children supported with the Cardiohelp ECMO System with the goal to plan a phase III (pivotal) randomized clinical trial

The main questions the Cardiohelp single-arm trial seeks to answer are:

* What is the safety and effectiveness of the Cardiohelp device for pediatric ECMO?
* Should the Cardiohelp device be FDA-cleared for children based on the results of the study?
* What are the optimal performance specifications of the Cardiohelp device in children?

The main questions the blood thinner randomized trial seeks to answer are:

* Which blood thinner is more promising (i.e., more effective and safer) in children on the Cardiohelp device?
* How should a pivotal trial of heparin vs. bivalirudin be designed so it is the most informative and efficient to determine the best blood thinner?

Children who are receiving the Cardiohelp device will be approached and consented to participate if interested. For the Cardiohelp device trial, participants will undergo a standardized data collection to estimate survival to 30 days and the prevalence of serious adverse events like stroke, bleeding, and hemolysis. For the blood thinner randomized trial, participants will be randomized 1:1 to blood thinner strategy to determine which blood thinner has the fewest bleeding and clotting complications.

For the Cardiohelp single-arm trial, participant outcomes will be compared to performance goals (PG) derived from the ECMO literature. For the blood thinner randomized trial, the amount of bleeding and clotting will be measured.

The study is funded by an R01 grant from the FDA's Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
This is a multicenter clinical trial to evaluate the safety and effectiveness of the Cardiohelp System for up to 30 days of support in children with severe cardiac failure. The trial includes a secondary randomized study comparing heparin versus bivalirudin anticoagulation according to standard treatment protocols.

Despite more than 50 years of ECMO use that carries up to 50% mortality, no standalone ECMO device has ever received FDA clearance for pediatric ECMO. All ECMO use in children is off-label, which may contribute to substantial mortality and complications, as well as wide center-to-center variation in ECMO practices that lacks an evidence base. Additionally, while two anticoagulants (heparin and bivalirudin) are commonly used in ECMO circuits, the optimal choice remains unknown-specifically, which anticoagulant is associated with the fewest circuit clots and least bleeding.

This study, funded by an R01 clinical trials Orphan Grant from the FDA, seeks to change the current status quo. By collecting systematic safety and effectiveness data on the Cardiohelp Device, we aim to determine whether it is safe and effective enough to become the first standalone ECMO device to receive FDA clearance for up to 30 days of support in children. The FDA clearance decision will be based on how the Cardiohelp performs relative to several key performance benchmarks drawn from the published ECMO literature, which the FDA has jointly agreed upon. These benchmarks include overall survival without severe stroke, degree of hemolysis (red blood cell breakdown), frequency of circuit change due to thrombus or device malfunction, stroke rate, and kidney injury rate.

For the anticoagulant randomized trial, we will collect systematic data on clotting and bleeding complications associated with each anticoagulant. As a Phase II study, the goal is not to reach a final answer, but to design a Phase III (pivotal) trial that is as informative and efficient as possible for addressing this critical question in the field of ECMO.

Tertiary goals of the study are: (1) to determine the optimal performance range (i.e., device specifications) for the Cardiohelp device in children to inform an eventual FDA label and Instructions for Use (IFU); and (2) to provide the FDA with a predicate device to support FDA clearance of other ECMO systems under 510(k) regulation, as no predicate devices currently exist to support such regulatory comparisons.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 to 16 years of age (i.e., <17 years)
2. Body weight 3 to 80 kilograms
3. VA-ECMO use for primary cardiac failure using the Cardiohelp system.
4. First ECMO run during the current hospitalization

Exclusion Criteria:Children must not meet any of the following exclusion criteria within 48 hours prior to device implant:

1. Gestationally-corrected age <37 weeks
2. Bleeding or coagulopathy that is a contraindication to anticoagulation
3. Irreversible renal, hepatic or lung failure
4. Stroke or uncertain neurological status within the past 30 days
5. Severely malnourished
6. Use of an ECMO system other than the Cardiohelp
7. VV-ECMO or ECMO for primary respiratory failure
8. Goals of patient to focus on comfort measures only.
9. Failure to separate from cardiopulmonary bypass
10. Allergy or contraindication to receiving UFH or bivalirudin as a primary anticoagulant on ECMO.
11. Patients who are pregnant or breastfeeding.
12. Unable to undergo randomization within 30 hours following ECMO cannulation (randomized cohort only)

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Survival to 30 days, recovery, ventricular assist device implant or transplant in the absence of severe symptomatic stroke (primary device effectiveness) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  Survival in the absence of severe symptomatic stroke to 30 days or decannulation for recovery, transplant or VAD implant. For patients with stroke definitely or probably related to ECMO, symptoms and severity will be determined at hospital discharge or 90 days, whichever is first.
Symptomatic stroke (primary device safety) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  For patients with stroke definitely or probably related to ECMO, the presence of stroke symptoms and its severity will be determined at hospital discharge or 90 days, whichever is first.
Severe hemolysis (primary device safety) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  Severe hemolysis as defined by the plasma-free hemoglobin level >100 mg/dL confirmed on repeat testing and outside the first 72 hours that is probably or definitely related to the device.
Circuit change due to thrombus (primary device safety) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  ECMO circuit change due primarily to thrombus that is probably or definitely related to the device.
Circuit change due primarily to device malfunction (primary device safety) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  Circuit change due primarily to device malfunction that is probably or definitely related to the device.
Renal injury/failure (primary device safety) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  renal injury/failure defined as three times the upper limit of normal or 3X baseline if the baseline is above the upper limit of normal.
Circuit-change free survival primarily due to thrombus (primary safety endpoint for anticoagulation RCT) | 30 days of ECMO support or ECMO explant, whichever is earlier.
  Circuit-change free survival where the circuit is change is primarily due to thrombus and is definitely or probably related to the anticoagulant (primary safety endpoint for anticoagulation RCT)
Bleeding | 30 days of ECMO support or ECMO explant, whichever is earlier.
  Total red blood cell transfusion volume in cc/kg/day probably or definitely related to the anticoagulant.

SECONDARY OUTCOMES:
Incidence of all serious adverse events | 30 days
  Incidence rate of all serious adverse events (per day of support)
NHLBI bleeding and clotting score | through 30 days of ECMO support or ECMO explant, whichever is earlier.
  The bleeding and clotting score as categorized by the ordinal 5-grade NHLBI score.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sleeper, ScD, Principal Investigator — Boston Children's Hospital; Caroline Ozment, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Cuimc/Nyph, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Children's Health Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No